CLINICAL TRIAL: NCT00528749
Title: Non-Invasive Measurement of Respiratory Effort
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Walter Reed Army Medical Center (U.S. Federal Agency)
Collaborators: Advanced Brain Monitoring, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: RespEffort
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2007-09-12 (Estimated); Status verified 2007-08

CONDITIONS: Upper Airway Resistance Syndrome
Keywords: Respiratory effort; Upper Airway Resistance Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Patient will wear ARES device while undergoing sleep study — Device is worn on forehead

SUMMARY:
This study is intended to compare intrathoracic pressure and respiratory effort data obtained by forehead venous pressure and respiratory movement (FVP/RM) with data obtained by the current gold standard, esophageal manometry. If this feasibility study validates the ability of FVP/RM data to quantitatively measure respiratory effort non-invasively, further studies will be performed to validate the utility of the ARES device in diagnosis of the UARS.

DETAILED DESCRIPTION:
Sleep apnea is the most common disorder observed in the practice of sleep medicine and is responsible for more morbidity and mortality than any other sleep disorder.(1) Although characterized over 40 years ago, sleep apnea has only recently gained recognition as one of the world's most prevalent undiagnosed disorders. Due to associated morbidity and mortality, sleep apnea has been identified as a major public health concern. Currently, sleep apnea is diagnosed by performing a sleep study. This requires a patient staying overnight in a sleep laboratory while being monitored, which is often inconvenient for patients and is relatively expensive to perform. The development of a device that allows for simple home monitoring of patients when assessing for sleep apnea would be a significant development in the field of sleep medicine.

The differentiation of obstructive sleep apnea (OSA) from central sleep apnea is an important aspect of diagnosing and treating OSA. In central apneas/hyponeas, the lack of airflow is due to lack of respiratory effort. In OSA, effort to breathe continues, but airflow is prevented by an occluded airway. More recently, subtle obstructive events without a defined desaturation, characterized by increasing respiratory efforts against a partially closed airway and terminated by an arousal, have been described as Upper Airway Resistance Syndrome (UARS). UARS can lead to daytime somnolence due to these frequent arousals. Although nasal pressure signal has been used as a surrogate, by definition, distinguishing UARS from OSA requires the use of esophageal manometry. This syndrome is characterized by increased upper airway resistance (IUAR) that was defined by increasingly negative inspiratory esophageal pressure. (2) To better understand the clinical significance of esophageal manometry, let us briefly review some basic physiology. Taking a breath requires that the inspiratory muscles generate sufficient force to overcome the elastic recoil of the chest wall and lungs, frictional lung and chest wall tissue resistance, and the frictional resistance of airflow through the airways. At the end of inspiration, the potential energy stored in the tissues of the lungs and chest wall is available to allow rapid passive exhalation when the inspiratory muscles cease contraction and the distending force disappears. All intrathoracic structures are subjected to the pressures generated by breathing. The esophagus is a thin walled muscular tube that, from the view of pulmonary physiologists, is ideally placed in the thoracic cavity between the lung surface and the chest wall. Measurement of differential pressure changes in the lumen of the esophagus accurately reflect changes in intrathoracic pressure. These changes in intrathoracic pressure are in turn reflective of inspiratory effort and have become the gold standard for detecting and quantifying inspiratory effort.

Unfortunately, measurement of esophageal manometry requires the placement of an esophageal catheter via the nose or mouth. This procedure in invasive, time consuming, and requires specialized training. For this reason, esophageal manometry is not routinely performed during sleep studies, although it is performed in patients at the WRAMC sleep lab who are suspected of having UARS. Instead of esophageal manometry, the most frequently used method of monitoring respiratory effort is to record thoracic cage expansion. In this procedure, bands are placed around the rib cage and abdomen. The change in circumference of these two compartments with breathing is measured. This procedure yields a qualitative change in inspiratory volume and paradoxical movement of the rib cage or abdomen can indicate effort against a closed or partially collapsed airway. This device is impractical for self-application by patients. Given the limitations of the latter procedure and the invasive nature of esophageal manometry, a non-invasive quantitative method for measuring respiratory effort would be a significant advancement in sleep medicine.

Over the past five years, investigators from Advanced Brain Monitoring, Inc. developed and validated the Apnea Risk Evaluation System (ARES). This device was initially developed to provide a highly accurate method of in-home diagnosis of OSA that maximized patient comfort and ease of use. The ARES Unicorder was designed as a single site (forehead) system to acquire oxygen saturation, pulse rate, snoring, airflow (nasal pressure), and head position/movement. Recently, investigators determined that a number of signals that were being acquired with the Unicorder could be used to measure respiration.(1) Pulsations observed in the red and infrared optical signals used to compute oxygen saturation and the forehead sensor pressure signal appear to reflect central venous pressure changes. These data has been termed the Forehead Venous Pressure/Respiratory Movement (FVP/RM) measure. If FVP/RM data proves to correlate with esophageal manometry data, the long sought after non-invasive quantitative measurement of intrathoracic pressure and respiratory effort would be available. This would represent a significant advancement in the diagnostic evaluation of sleep disordered breathing.

To better illustrate how forehead venous pressure could reflect intrathoracic pressure, let us again review some physiology. During inspiration, the central venous pressure (CVP) decreases, aiding the return of blood to the heart. Changes in pleural and intrathoracic pressure due to respiration are reflected by and can be timed to changes in central venous pressure. When recumbent, the internal and external jugular veins are open and provide the primary cerebral and superficial forehead venous return. The communication between the superior vena cava and the veins of the headallows intrathoracic pressure changes to be reflected by the superficial veins of the head. In a sense, the forehead veins offer a direct fluid filled catheter into the thoracic cavity, and when the correct compressive force is applied against the skull, respiratory effort linked venous pressure changes can be accurately measured.

In summary, current evaluation of UARS requires esophageal manometry testing, an invasive and time consuming procedure for accurate diagnosis. Currently, no non-invasive quanitative means of measuring intrathoracic pressure changes linked to respiratory effort exists. This study is a pilot trial of a new non-invasive method of determining intrathoracic pressures. If intrathoracic pressure data from this device is found to correlate with esophgeal manometry data, this could have significant implications on the way in which UARS is diagnosed. This technology also has the potential to develop a non-invasive means of measuring CVP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older,
* Referred for sleep study at WRAMC for suspected sleep disordered breathing.

Exclusion Criteria:

* Pregnancy
* Age <18
* Nasal defects precluding insertion of esophageal manometer
* Patients currently on anticoagulation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-02

PRIMARY OUTCOMES:
Comparison of respiratory effort data generated by esophageal manometer with that generated by ARES device | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed Army Medical Center, Washington D.C., District of Columbia, United States